CLINICAL TRIAL: NCT01192880
Title: A Phase III, Multi-Center, Randomized, 24 Week, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate Efficacy and Safety of RO4917838 in Stable Patients With Persistent, Predominant Negative Symptoms of Schizophrenia Treated With Antipsychotics Followed by a 28 Week, Double-Blind Treatment Period
Brief Title: A Study to Evaluate Efficacy and Safety of Bitopertin in Participants With Persistent, Predominant Negative Symptoms of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN25308; 2010-020470-42
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone; Antipsychotic Agents

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Bitopertin 10 mg + Antipsychotics (Experimental): Treatment Period 1: Participants will receive bitopertin 10 milligrams (mg) tablet orally once daily for 24 weeks. Treatment Period 2: Participants will receive bitopertin 10 mg tablet orally once daily for 28 weeks (up to Study Week 52). After Week 52 there will be a 4-week washout period for at least 50 percent (%) of participants (up to Week 56). Long-Term Extension: After Week 56, participants will enter the long term extension period and continue to receive bitopertin 10 mg tablet orally once daily up to 3 years. In addition, throughout the study, participants will continue their same stable antipsychotic treatment as they were receiving prior to entry in the study.
  Interventions: Drug: Bitopertin; Drug: Antipsychotics
- Bitopertin 20 mg + Antipsychotics (Experimental): Treatment Period 1: Participants will receive bitopertin 20 mg tablet orally once daily for 24 weeks. Treatment Period 2: Participants will receive bitopertin 20 mg tablet orally once daily for 28 weeks (up to Study Week 52). After Week 52 there will be a 4-week washout period for at least 50% of participants (up to Week 56). Long-Term Extension: After Week 56, participants will enter the long term extension period and continue to receive bitopertin 20 mg tablet orally once daily up to 3 years. In addition, throughout the study, participants will continue their same stable antipsychotic treatment as they were receiving prior to entry in the study.
  Interventions: Drug: Bitopertin; Drug: Antipsychotics
- Placebo (Placebo Comparator): Treatment Period 1: Participants will receive bitopertin matching placebo tablet orally once daily for 24 weeks. Treatment Period 2: Participants will receive bitopertin matching placebo tablet orally once daily for 32 weeks (up to Study Week 56). Long-Term Extension: After Week 56, participants will enter the long term extension period and will be switched to (in blinded manner) bitopertin 10 mg tablet orally once daily up to 3 years. In addition, throughout the study, participants will continue their same stable antipsychotic treatment as they were receiving prior to entry in the study.
  Interventions: Drug: Placebo; Drug: Antipsychotics

INTERVENTIONS:
Drug: Placebo — Participants will receive bitopertin matching placebo once daily for 56 weeks.
  Arms: Placebo
Drug: Bitopertin — Participants will receive 10 mg or 20 mg of bitopertin.
  Other Names: RO4917838
  Arms: Bitopertin 10 mg + Antipsychotics; Bitopertin 20 mg + Antipsychotics
Drug: Antipsychotics — Participants will continue to receive their stable antipsychotic regiment throughout the study. Study protocol does not specify any particular antipsychotic drug and regimen.

SUMMARY:
This Phase 3, multi-center, randomized, double blind, parallel-group, placebo-controlled study will evaluate the efficacy and safety of RO4917838 (bitopertin) in participants with persistent, predominant negative symptoms of schizophrenia. Participants, on stable treatment with antipsychotics, will be randomized to receive daily oral doses of RO4917838 or matching placebo for 52 weeks, followed by an optional treatment extension for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Based on the screening Structured Clinical Interview for and Statistical Manual of Mental Disorders, 4th Edition (DSM IV) - Clinical Trial (SCID CT), a DSM-IV- Text Revision (DSM-IV-TR) diagnosis of schizophrenia, paranoid, disorganized, residual, undifferentiated or catatonic subtype
* A score of 40 or greater on the sum of the 14 PANSS negative and disorganized thought factor items (items scored 1-7 for a maximum possible score of 98)
* A score of 22 or less on the sum of the 8 PANSS positive symptom factor items. The score of the items of P1 (delusions), P3 (hallucinatory behavior), P6 (suspiciousness) and G9 (unusual thought content) meet the following requirements: no more than 2 of the above items have a score of 4; all of the above items score less than 5
* Clinical stability for 6 months prior to randomization as well as antipsychotic treatment stability for the past 8 weeks at the time of randomization
* Are at least moderately ill, as defined by Clinical Global Impression - Severity (CGI S) of negative symptoms score more than or equal to (>/=) 4
* Stable doses of anticholinergic, antidepressive medication for at least 8 weeks prior to randomization is allowed as long as the respective scales cut-off entry criteria are met
* With the exception of clozapine, participants are on any of the available marketed atypical or typical antipsychotics (treatment with a maximum of 2 antipsychotics)
* Have a caregiver considered reliable by the investigator
* Female participants who are not either surgically sterile or post-menopausal must agree to use at least one effective forms of contraception from agree to remain sexually abstinent from screening until 90 days after the completion of the study medication

Exclusion Criteria:

* Evidence that participant has clinically significant, uncontrolled and unstable disorder (for example, cardiovascular, renal, hepatic disorder)
* Body Mass Index (BMI) of less than (<) 17 or more than (>) 40 kilograms per meter square (kg/m^2)
* Depressive symptoms, defined as a score of 9 or greater on the Calgary Depression Rating Scale for Schizophrenia (CDSS)
* A severity score of >/=3 on the Parkinsonism item of the Extrapyramidal Symptoms Rating Scale - Abbreviated (ESRS-A) (Clinical Global Impression, Parkinsonism)
* Positive result on the serum pregnancy test or are breast feeding at screening, or intend to become pregnant during the course of the trial.
* History of neuroleptic malignant syndrome (NMS)
* Based on the DSM-IV-TR criteria and screening SCID-CT have: other current DSM-IV-TR Axis I diagnosis; alcohol or substance dependence within 12 months or abuse within 3 months with the exception of nicotine; dementia, delirium and other amnestic disorder per DSM-IV-TR
* Treated with electroconvulsive therapy (ECT) within 6 months prior to randomization
* Ever received RO4917838 or another glycine transporter 1 (GLYT 1) inhibitor
* Require high doses of benzodiazepines (> 4 mg per day lorazepam or equivalent)
* Have a positive urine drug screen for amphetamines (including 3,4-Methylenedioxymethamphetamine [MDMA]/ecstasy), cocaine, barbiturate, cannabis and/or opiates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2010-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Mean Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Negative Symptom Factor Score at Week 24 | Baseline, Week 24
Percentage of Participants with Adverse Events | From baseline up to 24 weeks

SECONDARY OUTCOMES:
Mean Change from Baseline in the Personal and Social Performance (PSP) Total Score at Week 24 | Baseline, Week 24
Mean Change from Baseline in the PANSS Total Score at Week 24 | Baseline, Week 24
Mean Change from Baseline in the PANSS Factor Scores at Week 24 | Baseline, Week 24
Mean Change from Baseline in the PANSS Subscale Scores at Week 24 | Baseline, Week 24
Percentage of Participants With Response, as Assessed by PANSS Negative Symptom Factor Score | Week 24
Percentage of Participants with Response, as Assessed by CGI-I Overall and Negative Symptoms Rating Score | Week 24
Percentage of Participants with Both At Least 20% Improvement from Baseline in the PANSS Negative Symptom Factor Score and with a CGI-I Negative Symptoms Rating of Either Much or Very Much Improvement | Week 24
Mean Change from Baseline in the CGI-S Overall and Negative Symptoms Rating Score | Baseline, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (103):
- United States (27):
  - Clinical Innovtions Inc, Costa Mesa, California
  - Synergy Clinical Research of Escondido, Escondido, California
  - San Fernando Mental Health Center, Granada Hills, California
  - University of California San Diego, La Jolla, California
  - Excell Research, Oceanside, California
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - Collaborative Neuroscience Network Inc., Torrance, California
  - Behavioral Clinical Research Inc., Lauderhill, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Berma Research Group, Plantation, Florida
  - Atlanta Center For Medical Research, Atlanta, Georgia
  - Indiana University; LaRue Carter Memorial Hospital-Research Unit, Indianapolis, Indiana
  - Clinical Insights, Inc., Glen Burnie, Maryland
  - Precise Research Centers, Flowood, Mississippi
  - Altea Research Institute, Las Vegas, Nevada
  - Ocean Rheumatology, Toms River, New Jersey
  - State University of New York at Buffalo; Department of Psychiatry, Buffalo, New York
  - New York State Psychiatric Institute; Psychiatry Dept of Columbia University, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Duke University, Durham, North Carolina
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - Scranton Medical Institutes Llc., Scranton, Pennsylvania
  - Community Clinical Research Inc., Austin, Texas
  - University Hills Clinical Research, Irving, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Eastside Therapeutic Resource, Kirkland, Washington
- Bulgaria (8):
  - DDPDS Prof Dr Ivan Temkov EOOD, Burgas
  - MHAT Dr.Hristo Stambolski EOOD; Psychiatry Ward of Acute Psychotic Disiorders in Severe Stage, Kazanlak
  - State Psychiatric Hospital Sv. Ivan Rilski Novi Iskar; First Man Dept. and First Woman Dept., Novi Iskar
  - State Psychiatric Hospital - Pazardzhik AD; Department for active treatment of men and for women, Pazardzhik
  - UMHAT Dr Georgi Stranski; EAD; Psychiatry, Plovdiv
  - State Psychiatric Hospital Dr. G. Kissiov; 3-d Women Ward 1-st Men Ward, Radnevo
  - DDPDIU-Ruse; Men acute department Women acute department, Rousse
  - Military Medical Academy- MHAT, Sofia
- China (18):
  - Hebei Mental Health Centre, Baoding
  - Beijing Huilongguan Hospital; Department of Psychiatric, Beijing
  - Peking University Sixth Hospital; Department of Psychiatry, Beijing
  - Beijing An Ding Hosp.Capital Medical University; 5th Clinical Dept Depression Centre, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Guangzhou Brain Hospital, GuangzhouGuangdong
  - The First Affiliated Hospital of College of Medicine, Zhejiang University(First Hospital of Zhejiang, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University College, Hangzhou
  - The First Affilliated Hospital of Kunming Medical College, Kunming
  - Nanjing Brain Hospital, Nanjing
  - Shanghai Mental Health Center, Shanghai
  - Tongji Hospital of Tongji University, Shanghai
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi Mental Health Center, Wuxi
  - The First Affiliated Hospital of The Fourth Military Medical University (Xijing Hospital), Xi'an
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Xi'an Mental Health Center, Xi'an
- Czechia (8):
  - Saint Anne s.r.o., Brno
  - Krajska nemocnice Liberec a.s., Liberec
  - Psychiatricka ambulance, Mělník
  - A-Shine s.r.o., Pilsen
  - Clintrial,s.r.o., Prague
  - Medical Services Prague s.r.o., Prague
  - Psychiatricke Centrum Praha, Praha 8 - Bohnice
  - CTCenter MaVe s.r.o., Sternberk
- Italy (8):
  - Azienda Ospedaliero-Universitaria Consorziale Pol. di Bari; Neuroscienze e Organi di Senso, Bari, Apulia
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Asst Degli Spedali Civili Di Brescia; Servizio di farmacia, Brescia, Lombardy
  - Clinica Mangiagalli, Milan, Lombardy
  - ASST FATEBENEFRATELLI SACCO; Psichiatria (Fatebenefratelli), Milan, Lombardy
  - Azienda Ospedaliero Universitaria Molinette San Giovanni Bat, Turin, Piedmont
  - A.O. Universitaria Pisana; Psichiatria, Pisa, Tuscany
  - Azienda Ospedaliera di Padova, Padua, Veneto
- Japan (26):
  - Kohnodai Hp., National Center for Global Health and Medicine, Chiba
  - Fukkokai Soubu Hospital, Funabashi-shi
  - Daiwakai Seimou Hospital, Gunma
  - Koseikai Kusatsu Hospital, Hiroshima
  - Hokkaido University Hospital, Hokkaido
  - NHO Hizen Psychiatric Medical Center, Kanzaki-gun
  - Sankeikai Nishigahara Hospital, Kita-ku
  - Hospital of the University of Occupational and Environmental Health,Japan, Kitakyushu-shi
  - Jinseikai Hosogi Unity Hospital, Kochi
  - NHO Kikuchi National Hospital, Koshi-shi
  - Yuge Hospital, Kumamoto
  - Jinkokai Kurayoshi Hospital, Kurayoshi-shi
  - NHO Higashiowari Hospital, Nagoya
  - Shinkokai Shiranui Hospital, Omuta-shi
  - Asakayama General Hospital, Sakaishi
  - Tonankai Ashirbetsu Hospital, Sapporo
  - Sawayamakai Teine Hospital, Sapporo
  - Tohoku Seishin Hokenkai Aoba Hospital, Sendai
  - Jisenkai Nanko Psychiatric Institute, Shirakawa-shi
  - Tokyo Women's Medical University Hospital, Tokyo
  - National Center Of Neurology And Psychiatry Hospital, Tokyo
  - Korenkai Minamitoyama Nakagawa Hospital, Toyama
  - Fujita Health University Hospital, Toyoake-shi
  - Deep Intention Hiyoshi Hospital, Yokohama
  - Kanagawa Prefectural Psychiatric Center Kinko Hospital, Yokohama
  - Yokohama Aihara Hospital, Yokohama
- Russia (8):
  - Kemerovo Regional Clinical Psychiatric Hospital, Kemerovo
  - GUZ Lipetsk Regional psychoneurological Hospital #1; Dispansary Department, Lipetsk
  - Institution of RAMS (Mental Health Research Center of RAMS); Psychopharmacology laboratory, Moscow
  - Central Moscow Regional Clinical Psychiatric Hospital, Moscow
  - City Psychiatric Hospital #2 of St. Nikolay Chudotvorets, Saint Petersburg
  - StP SR Psychoneurological Institute n.a.V.M.Bekhterev of MoH, Saint Petersburg
  - MHI City Clinical Hospital #2 named after V.I. Razumovsky; Psychiatric, Sartatov
  - Arkhangelsk Regional Clinical Psychiatric Hospital, Talagi

REFERENCES:
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500
- [Derived] Bugarski-Kirola D, Blaettler T, Arango C, Fleischhacker WW, Garibaldi G, Wang A, Dixon M, Bressan RA, Nasrallah H, Lawrie S, Napieralski J, Ochi-Lohmann T, Reid C, Marder SR. Bitopertin in Negative Symptoms of Schizophrenia-Results From the Phase III FlashLyte and DayLyte Studies. Biol Psychiatry. 2017 Jul 1;82(1):8-16. doi: 10.1016/j.biopsych.2016.11.014. Epub 2016 Dec 15. PMID 28117049